CLINICAL TRIAL: NCT02758600
Title: Cardiopulmonary and Metabolic Responses in Early Exercise-based Rehabilitation in Patients With or Without Left Ventricular Dysfunction After Coronary Arterial Bypass Grafting
Brief Title: Cardiopulmonary and Metabolic Responses to Early Exercise in Patients After Coronary Arterial Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Isadora Salvador Rocco, Principal Investigator, Federal University of São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 53016216.3.0000.5505
Record Dates: First submitted 2016-04-23; First posted 2016-05-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Acute Myocardial Infarction: Rehabilitation Phase; Coronary Artery Bypass Graft Triple Vessel; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LVEF < 45% (Experimental): Patients with left ventricular dysfunction will be evaluated before and 6 days after after coronary arterial bypass graft surgery. Postoperatively, subjects will be submitted to a portable cycle ergometer exercise protocol from the first day until hospital discharge.
  Interventions: Other: Cycle ergometer exercise rehabilitation protocol
- LVEF > 45% (Experimental): Patients without left ventricular dysfunction will be evaluated before and 6 days after after coronary arterial bypass graft surgery. Postoperatively, subjects will be submitted to a portable cycle ergometer exercise protocol from the first day until hospital discharge.
  Interventions: Other: Cycle ergometer exercise rehabilitation protocol

INTERVENTIONS:
Other: Cycle ergometer exercise rehabilitation protocol — Patients will be submitted to a progressive and moderate exercise protocol with a portable cycle ergometer.

SUMMARY:
Coronary arterial bypass graft surgery (CABG) is proven safe with improved survival and greater quality of life in patients with coronary arterial disease. Evidences on the cardiovascular and gas-exchanges responses during and right after early exercise-based rehabilitation of this patients are limited. Objective: The investigators aim to analyse breath-by-breath cardiopulmonary and metabolic responses during six-minute walk test (6MWT) and shuttle walk test (SWT) in patients with or without left ventricular dysfunction (LVD) after CABG. In addition, the investigators will investigate oxygen consumption and cardiopulmonary responses during the early exercise-based rehabilitation in the first days after surgery. Methods: According to the left ventricular ejection fraction (LVEF), subjects will be allocated into two groups: with LVD (LVEF < 45%) and without LVD (LVEF > 45%). Patients will be submitted to the 6MWT and SWT linked to portable spirometric-telemetric device before and 6 days after CABG. During the first days after surgery, patients will be evaluated about pulmonary function and respiratory strenght at rest and oxygen consumption during the portable cycle ergometer protocol. Clinical outcomes as time to hospital discharge, pulmonary complications and occurence of arrythmias will be assessed during inpatient time until hospital discharge. Incidence of mortality, hospital readmission and angina recurrence will be evaluated in a one-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 to 75 years old;
* Coronary arterial disease proved by coronary angiography
* Elective Coronary arterial bypass grafting

Exclusion Criteria:

* Pulmonary chronic disease
* Disabling neurological or orthopedic disease
* Morbidity obesity
* Urgency surgery
* Bilateral pleural opening
* Arrhythmias during exercise protocol
* Prolonged mechanical ventilation (>12 hours)
* Inability to comprehend or perform the tests

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test to measure functional capacity | 6 days
  According to the preoperative six-minute walk test linked to portable ergoespirometry device, we will evaluate the decrease in functional capacity in the sixth day after surgery.
Short-term complications | Until hospital discharge, an average of 15 days
  Incidence of arrythmias, pulmonary complications (pleural effusion, pulmonary atelectasis and pneumonia)
Shuttle walk test to measure functional capacity | 6 days
  According to the preoperative shuttle walk test linked to portable ergoespirometry device, we will evaluate the decrease in functional capacity in the sixth day after surgery.

SECONDARY OUTCOMES:
Pulmonary Dysfunction | 6 days (on the 1th, 3th and 6th day after surgery)
  By spirometry, assessing the decrease in forced vital capacity and changes in exhaled volume forced in first second postoperativetly compare to preoperative period.
Respiratory weakness | 6 days (on the 1th, 3th and 6th day after surgery)
  By manovacuometry, assessing the change in inspiratory muscle pressure and expiratory muscle pressure postoperativetly compare to preoperative period.
Oxygen Consumption | First 6 days after surgery
  Evaluate the oxygen consumption in metabolic equivalents (METS) during the cycle ergometer in post operative period by using spirometic-telemetric portable device during sessions.
Mid and Long Term Complications | 3 months to 1 year
  Complications such as angina recurrence, hospital readmission, cardiac events and all cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitary Hospital of Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No